CLINICAL TRIAL: NCT01894503
Title: A Clinical Evaluation of the Safety and Performance of the Steroid-Releasing S8 Sinus Implant When Used in Post-Sinus Surgery Patients With Recurrent Sinus Polyps
Brief Title: Safety and Performance of the Steroid-Releasing S8 Sinus Implant
Acronym: S8PK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P500-0513
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-03

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Bilateral in-office placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S8 Sinus Implant (Experimental): Bilateral in-office placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Interventions: Drug: S8 Sinus Implant (mometasone furoate, 1350 mcg)

INTERVENTIONS:
Drug: S8 Sinus Implant (mometasone furoate, 1350 mcg) — Bioabsorbable sinus implant with 1350 mcg of mometasone furoate released over 90 days
  Other Names: SINUVA (mometasone furoate) sinus implant

SUMMARY:
The purpose of this study was to assess the safety and performance of the steroid-releasing S8 Sinus Implant when used in post-sinus surgery patients who presented with recurrent sinus obstruction.

DETAILED DESCRIPTION:
The S8 PK study was a single-center, open label study treating 5 adult (18 years or older) patients diagnosed with chronic sinusitis, who had undergone prior bilateral total ethmoidectomy and later presented with recurrent nasal obstruction/congestion symptoms and bilateral ethmoid polyposis. The S8 PK study assessed the safety, implant delivery to the ethmoid sinus, and systemic exposure to mometasone furoate (MF) by measuring plasma MF and cortisol concentrations through 30 days post-procedure.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older
* Diagnosis of chronic sinusitis
* Prior bilateral total ethmoidectomy
* Recurrent sinus obstruction due to polyps grade 2 or higher

Key Exclusion Criteria:

* Required use of mometasone furoate within 2 weeks prior to implant procedure
* Significant scarring or adhesions of the sinus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Ow, MD, Principal Investigator — Sacramento ENT
Locations (1):
- Sacramento ENT, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective, single-center open label study treating adult patients with recurrent polyposis after bilateral total ethmoidectomy. Study period 9 July 2013 to 17 July 2013
Pre-assignment Details: A total of six patients were enrolled (consented). One patient did not have the required grade 2 polyposis on at least one ethmoid side and was excluded. The remaining five patients meet all eligibility criteria and underwent an in-office bilateral placement of two S8 Sinus Implants. All five patients completed follow-up through the Day 90 visit.
Groups:
- S8 Sinus Implant: Bilateral in-office placement of the S8 Sinus Implant (mometasone furoate sinus implant, 1350 mcg) in the ethmoid sinuses S8 Sinus Implant (mometasone furoate, 1350 mcg): Bioabsorbable sinus implant with 1350 mcg of mometasone furoate released over 90 days
Period: Overall Study
Arm/Group | S8 Sinus Implant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Demographic and Baseline Clinical Characteristics: In-office bilateral placement of two S8 Sinus Implants
Arm/Group | Demographic and Baseline Clinical Characteristics
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 46.2 [37 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Sinuses With Successful Implant Delivery
Description: Defined as successful access and deployment of the S8 Sinus Implant to the target ethmoid sinus at the end of the baseline procedure
Time Frame: End of baseline procedure
Population: Per-treatment evaluable population, consisting of all sinuses in which placement of the S8 Sinus Implant was attempted.
Measure: Count of Units; unit: Sinuses
Units Other Than Participants: Sinuses
Groups:
- S8 Sinus Implant: Implant delivery success
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 5
Number analyzed (Sinuses) | 10
Sinuses | 10

2. Secondary Outcome: Number of Patients With Plasma Mometasone Furoate Concentration >LLOQ
Description: Concentration of mometasone furoate was determined in blood samples collected at baseline, Days 3, 7, 14, 21 and 30 using a validated method with the lowest level of quantification (LLOQ) of 30 pg/ml.
Time Frame: Days 3, 7, 14, 21 and 30
Population: Per-treatment evaluable population consisting of all patients
Measure: Number; unit: participants
Groups:
- S8 Sinus Implant: In-office bilateral placement of the S8 Sinus Implant (1350 mcg of mometasone furoate) in the ethmoid sinuses
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 5
participants
  Baseline | 0
  Day 3 | 3
  Day 7 | 1
  Day 14 | 2
  Day 21 | 0
  Day 30 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were recorded and tabulated through Day 90.
Arm/Group | S8 Sinus Implant
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S8 Sinus Implant (N=5)
Headache (Nervous system disorders) | 1 (1) — Mild
Acute sinusitis (Infections and infestations) | 1 (1) — Mild, maxillary sinus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is NOT an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.